CLINICAL TRIAL: NCT06454136
Title: A Randomized Controlled Pilot Trial of Mobile Technology for Reducing and Preventing Adolescent Suicidality
Brief Title: Pilot Trial of Mobile Technology for Adolescent Suicidality
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oui Therapeutics, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-Oui-001; 6R42MH125691-03 (NIH)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: OTX-207
- Control (Sham Comparator)
  Interventions: Device: Comparator App + Treatment as Usual (TAU)

INTERVENTIONS:
Device: OTX-207 — Experimental Pscyhoeducation and Intervention App
  Arms: Treatment
Device: Comparator App + Treatment as Usual (TAU) — Digitized content and information included in standard of care (i.e., TAU)
  Arms: Control

SUMMARY:
The primary objective of this study is to assess the efficacy of a digital intervention in reducing suicidal ideation in adolescents.

DETAILED DESCRIPTION:
This double blind, randomized controlled trial will evaluate the preliminary efficacy of two digital interventions among 114 adolescent participants, and their parents/guardians, in reducing suicidal ideation in the adolescent participants. Adolescent participants, parent/guardian participants, and research assessors will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (of any sex), ages 13 to 17 years
2. Patients who were recently hospitalized and have:

   1. attempted suicide or
   2. have documented SI and a history of attempted suicide, as verified by the Columbia-Suicide Severity Rating Scale (C-SSRS).

   Hospitalized is defined as admission to a medical or psychiatric service for further assessment and care including observation units, intensive care or other medical units and psychiatric units.
3. Patient owns a smartphone capable of downloading and running apps
4. Patient is willing and able to complete enrollment procedures
5. Patient and Parent/Guardian are willing to assent/consent to medical record review for one year following randomization to collect suicide attempt data
6. Patient and Parent/Guardian are able to understand the nature of the study and sign documentation of written informed assent (Patient) and consent (Parent/Guardian)
7. Patient and Parent/Guardian understand written and spoken English
8. Patient is willing to agree to release of information to their Parent/Guardian and providers when clinically indicated

Exclusion Criteria:

1. Patients who are acutely intoxicated or in detoxification at the time of enrollment
2. Patients who are currently enrolled in other treatment studies for the symptoms and behaviors targeted
3. Patients who are incapable of understanding and following through with the study procedures (e.g., cognitive impairment)
4. Patients with a psychiatric or medical condition or custody arrangement that, in the opinion of the PI, may compromise, interfere, limit, affect or reduce the patient's ability to provide informed consent, complete the study, or may adversely impact the safety of the patient or the integrity of the data. Examples of considerations include terminal illness where death would be anticipated before completing study procedures, active psychosis at the time of assent, severe or unstable medical condition.
5. Patients whose discharge plans include transfer to inpatient care, as confirmed by the index hospitalization discharge summary/plan.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicide Ideation (SSI) | 12 weeks
  Change in suicidal ideation between baseline and 12 weeks after randomization will be assessed using the Scale for Suicide Ideation (SSI) most severe point of illness score. The possible range of scores is 0-38, where a higher score indicates greater severity of suicide ideation.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hartford HealthCare, Hartford, Connecticut
  - University of Cincinnati, Cincinnati, Ohio
  - Rhode Island/Bradley Hospital/Brown Health University, Providence, Rhode Island